CLINICAL TRIAL: NCT04423978
Title: Implications of Covid-19 on the Lifestyle Changes and Supports Used (ICOLS): a Survey in the Province of Reggio Emilia
Brief Title: Implications of Covid-19 on the Lifestyle Changes
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: ICOLS_CovidStyle
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: Italy; Lifestyle; Pandemics; Quarantine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Northern Italy has been profoundly touched by the Covid-19 pandemic. To limit the outbreaks of contagion, the Italian government imposed 2.months of complete lock-down, which imposed the social isolation for the whole population and, for those positive to the Covid-19, the complete confinement at home. Despite the recommendations for conserving healthy lifestyle of the Italian Government, during the lock-down the likelihood to fall into unhealthy behaviours might have increased.

This study aims to describe the impact of Covid-19 on the lifestyles of a population of Italian adults living in an area of high spread of Sars-CoV-2.

DETAILED DESCRIPTION:
The aims of this study were to detect the changes in lifestyles occurred during the imposed lock-down phase and the support services used the most by participants.

This study consists in the administration of an on-line survey addressed to adult individuals living in the province of Reggio Emilia (Italy). The survey was posted on-line on the website of the Azienda USL- IRCCS di Reggio Emilia and it was spread to the community through apps and social networks.

The on-line survey is free to access, self-administered and it consists of 50 questions. The questions investigates the changes occurred in employment status, physical exercise, diet, tobacco and alcohol consumption, sleep quality and leisure activities during the pandemic lock-down phase as well as the available local support services used and perceived as useful.

ELIGIBILITY:
Inclusion Criteria:

* adult individuals living in the province of Reggio Emilia (Italy)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study aims to describe the impact of Covid-19 on the lifestyles of a population of Italian adults living in the province of Reggio Emilia (Italy), an area of high spread of Sars-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 1826 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
The ratio of individuals living in the province of Reggio Emilia who completed the survey | 1 month and a half
  We will report the number of inhabitants of the Province of Reggio Emilia who answered the survey

SECONDARY OUTCOMES:
The ratio of individuals who changed the lifestyles during the lock-down | 1 month and a half
  We will report the number of inhabitants of the Province of Reggio Emilia who changed their lifestyles during the lock-down phase
The number and the type of support services used the most by participants | 1 month and a half
  We will report the number of inhabitants of the Province of Reggio Emilia who used and appreciated the supprt services to overcome the lock-down phase

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mazzini, MD, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (1):
- Elisa Mazzini, Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No